CLINICAL TRIAL: NCT06520761
Title: The Effect of Injectable Platelet Rich Fibrin Versus Low-Level LASER Therapy on The Rate of Orthodontic Tooth Movement
Brief Title: The Effect of Injectable PRF Vs LLL on Orthodontic Tooth Movement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Faculty of Dental Medicine for Girls (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: ORTHO-108-5-b
Record Dates: First submitted 2024-07-20; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2023-10

CONDITIONS: Rate of Canine Retraction; Root Resorption
MeSH Terms: conditions — Root Resorption | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- injectable platelet rich fibrin (Experimental): blood sample is collected from the patient, centrifuged at 700rpm for 3 minutes then the resulted injectable platelet rich fibrin is injected around the upper right canine while the upper left canine act as a control
  Interventions: Procedure: Injectable platelet rich fibrin
- Low Level LASER (Experimental): low level laser from diode laser machine is applied around the upper right canine and the upper left canine acts as a control
  Interventions: Device: Low Level LASER

INTERVENTIONS:
Procedure: Injectable platelet rich fibrin — blood sample obtained from the participant, centrifuged at 700 rpm to produce injectable platelet rich fibrin, this will be injected around the upper canine
  Arms: injectable platelet rich fibrin
Device: Low Level LASER — Diode LASER device is used to apply Low Level LASER around the upper canine
  Arms: Low Level LASER

SUMMARY:
The purpose of the present study is to compare the effect of injectable platelet fibrin and Low Level LASER therapy on the rate of upper canine retraction, and on root resorption of the canine

DETAILED DESCRIPTION:
the study involves two groups the first group received low level laser at the upper right canine, while the upper left canine act as a control. The second group received injectable platelet rich fibrin at the upper right canine, while the upper left canine act as a control. in each group we will compare rate of canine retraction between both sides, and amount of root resorption also we will compare both groups regarding rate of canine retraction and amount of root resorption

ELIGIBILITY:
Inclusion Criteria:

1. Patients with age 18 years or older.
2. Presence of all permanent teeth except for the third molar.
3. Presence of malocclusion requiring maxillary first premolar extraction such as (class II division 1 or bimaxillary dentoalveolar protrusion).

Exclusion Criteria:

1. Patient with a history of previous orthodontic treatment.
2. Medical problems may interfere with orthodontic treatment.
3. Bad oral hygiene.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Rate of canine retraction | 4 month
  measure the rate of distal movement of the upper canine

SECONDARY OUTCOMES:
Root resorption of upper canine | 4 month
  measure root resorption of upper canine

CONTACTS AND LOCATIONS:
Overall Officials: Samir A Ebrahim, Professor, Principal Investigator — Head of orthodontic department at faculty of Dental Medicine for Girls Al-Azhar university
Locations (1):
- Faculty of Dental Medicine for Girls Al Azhar university, Cairo, Naser City, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zeitounlouian TS, Zeno KG, Brad BA, Haddad RA. Effect of injectable platelet-rich fibrin (i-PRF) in accelerating orthodontic tooth movement : A randomized split-mouth-controlled trial. J Orofac Orthop. 2021 Jul;82(4):268-277. doi: 10.1007/s00056-020-00275-x. Epub 2021 Jan 22. PMID 33481053
- See also: The role of platelet-rich fibrin (PRF) in accelerating orthodontic tooth movement has been controversially discussed in available clinical studies. Objective: To investigate the effectiveness of i-PRF in accelerating maxillary canine retraction. — https://pubmed.ncbi.nlm.nih.gov/33481053/